CLINICAL TRIAL: NCT07404644
Title: Vonvendi Intravenous Specified Drug Use-results Survey "Pediatric Administration"
Brief Title: An Observational Study of Vonicog Alfa (rVWF) in Pediatric Participants With Von Willebrand Disease (vWD)
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-577-4010
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Von Willebrand Disease (vWD)
Keywords: Von Willebrand Disease (vWD)
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- vonicog alfa (rVWF) Group: Participants with Von Willebrand Disease (vWD) who received vonicog alfa (rVWF) in accordance with package insert.
  Interventions: Drug: vonicog alfa (rVWF)

INTERVENTIONS:
Drug: vonicog alfa (rVWF) — rVWF administered by intravenous injection.
  Other Names: Vonvendi Intravenous; Recombinant von Willebrand Factor (rVWF); TAK-577

SUMMARY:
This study is conducted in Japan of vonicog alfa (rVWF) used to treat pediatric participants with Von Willebrand Disease (vWD).

The main aim of the study is to evaluate adverse drug reaction and effectiveness of vonicog alfa (rVWF).

During the study, pediatric participants with vWD will be administered with rVWF under routine normal practice. The investigators will evaluate adverse events due to rVWF for 1 year from the start of drug administration.

The study sponsor will not be involved in how the participants are administered but will be recorded what happens during the study.

ELIGIBILITY:
Inclusion Criteria :

* Under 18 years old with vWD.
* Participants who are treated with rVWF for the purpose of hemostatic treatment and management during bleeding episodes or perioperative periods.
* Participants who have prescription or administration after the approval date of rVWF for pediatric use in Japan.

Exclusion Criteria :

- Patients who are participating in clinical trials of rVWF.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The population of this study are all participants who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2031-05-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience at Least One Adverse Drug Reactions (ADRs) | Up to 1 year
  Adverse Event (AE) refers to any undesirable medical occurrence in a patient administered a drug, regardless of causal relationship. This includes any unfavorable or unintended sign (including abnormal laboratory findings), symptom, or disease occurring during administration, regardless of causal relationship. Adverse drug reaction (ADR) refers to AE related to administered drug.

SECONDARY OUTCOMES:
Hemostatic Efficacy Assessed by Hemostatic Efficacy Rating Scale | 1 year
  Hemostatic efficacy for bleeding episodes will be assessed by a predefined 4-point rating scale (Excellent, Good, Moderate, None).
Hemostatic Efficacy during Perioperative Periods Assessed by Hemostatic Efficacy Rating Scale | 1 year
  Hemostatic efficacy during perioperative periods will be assessed by a predefined 4-point rating scale (Excellent, Good, Moderate, None).
Number of Infusions per Bleeding Episode | 1 year
Number of Infusions during Perioperative Periods | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).